CLINICAL TRIAL: NCT03901677
Title: Effects of Tai Chi Exercise on Balance and Body Awareness of Younger Adults
Brief Title: Tai Chi Exercise on Balance and Awereeness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ayça Aytar TIĞLI, Principal Investigator, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA19/10
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2019-04

CONDITIONS: Young Adult
Keywords: exercise; Awareness; posture
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Masking Description: All assessments done by masked therapist to avoid bias who have no idea about intervention before and 12 weeks after the tai chi exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai-chi training (Experimental): Tai-chi training performe as a group exercise. Duration for tai chi exercise will be 60 minutes for 2 days per week for 12 weeks. Each session includes 10 min warm-up and cool-down and 40 min Tai Chi exercises. During exercises, attention paid to correct positioning of the upper and lower extremity joints, and mentally concentration achieve. Slow and controlled movements will carry out by a specialized physiotherapist.
  Interventions: Other: Tai-chi training

INTERVENTIONS:
Other: Tai-chi training — Group exercise apply with physiotherapist

SUMMARY:
The aim of this study is to determine the effect of Tai chi exercises on balance and body awareness in younger adults. Forty-two healthy subjects between the ages of 18-25 who do not have any restriction to exercise participate in our study. After recording the sociodemographic characteristics of the subjects, static and dynamic balance and body awareness will be evaluated. Kinesthetic Ability Trainer will be used to assess static and dynamic balance and body awareness will be evulated with Body Awareness Questionnaire. All assessments will be done before and 12 weeks after the tai chi exercise. Tai-chi training will be performed as a group exercise. Duration for tai chi exercise will be 60 minutes for 2 days per week totally 12 weeks.

DETAILED DESCRIPTION:
Tai-chi training was performed as a group exercise. Duration for tai chi exercise was 60 minutes for 2 days per week for 12 weeks. Each session includes 10 min warm-up and cool-down and 40 min Tai Chi exercises. During exercises, attention was paid to correct positioning of the upper and lower extremity joints, and mentally concentration was achieved. Slow and controlled movements were carried out by a specialized physiotherapist

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 18-25,
2. Subjects who had lack of disease.

Exclusion Criteria:

1. Subjects with neurological symptoms,
2. Subjects with orthopedic problems,
3. Subjects with heart failure,
4. Subjects with respiratory distress.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Body Awareness Questionnaire | 12 week
  Body awareness will be evaluated with Body Awareness Questionnaire (BAQ). It is a questionnaire composed of 4 subgroups (changes in the body process, sleep-wake cycle, estimation of the onset of the disease, estimation of the body reactions) and a total of 18 expressions to determine the normal or non-normal sensitivity level of the body composition. Subjects assess each item from 1 to 7. Higher scores on the BAQ indicates higher awareness.

SECONDARY OUTCOMES:
Balance Test | 12 week
  Kinesthetic Ability Trainer (KAT) 3000 (KAT 3000, Berg, Vista, CA, USA) will be used to assess static and dynamic balance. The KAT 3000 consists of a movable platform supported on a central point by a small pivot. A tilt sensor on the platform is connected to a computer, which registers the deviation of the platform from a reference position 18.2 times each second. The distance from the central point to the reference position is measured at every registration. From the summation of these distances, a score, the balance index (BI), can be calculated (a low BI implies good ability to perform the balance test).

CONTACTS AND LOCATIONS:
Overall Officials: ayca tigli, Phd, Principal Investigator — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No